CLINICAL TRIAL: NCT01370486
Title: Double Blind, Randomised, Cross-over Study Melatonin Versus Placebo in the Lennox-Gastaut Syndrome: Neurophysiological and Neuropsychological Effects
Brief Title: Melatonin Versus Placebo in the Lennox-Gastaut Syndrome: Neurophysiological and Neuropsychological Effects
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study did not received the approbation from Swissmedic. Therefore, the recruitment of participants never started.
Sponsor: Institution de Lavigny (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25/10
Record Dates: First submitted 2011-06-08; First posted 2011-06-10 (Estimated); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Lennox-Gastaut Syndrome
Keywords: Lennox-Gastaut syndrome; Epileptic encephalopathy; Melatonin; Tonic seizures; Interictal discharges; Quality of sleep
MeSH Terms: conditions — Lennox Gastaut Syndrome; Seizures; Sleep Initiation and Maintenance Disorders | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- melatonin (Active Comparator)
  Interventions: Drug: melatonin
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: melatonin — melatonin cp 2 mg 1x/d for 1 month
  Other Names: brand name: circadin
  Arms: melatonin
Drug: placebo — placebo cp 1x/d for 1 month
  Arms: placebo

SUMMARY:
Lennox-Gastaut syndrome is a severe epileptic encephalopathy of childhood. In that syndrome, various type of seizure occur, mainly tonic seizures, atonic seizures and atypical absences. The tonic seizure occur mostly at night.

The hypothesis is that the melatonin could have a positive effect in that syndrome, by reducing the epileptic activity (assessed in the polysomnographic record by counting the number of interictal and ictal discharges) and stabilizing the structure of sleep.

The study is double blind, randomised, cross-over designed.

DETAILED DESCRIPTION:
The aim of the trial is to study the efficacity of melatonin in the Lennox-Gastaut syndrome, by assessing the reduction of the seizure/interictal discharges in polysomnography and assessing the sleep structure.

After initial recruitment, the baseline visit includes a polysomnography. The patients will then be randomised in two groups: melatonin (1 cp containing melatonin 2 mg 1x/d 1h before sleep) vs placebo (1 cp 1x/d 1h before sleep). The treatment (melatonin or placebo) will be given for 1 month.

After 1 month, the treatment will be stopped and another polysomnography will be recorded.

The patients will take no treatment (wash-out period) for 15 days. The second treatment phase is cross-over: the group that had melatonin in the first phase will take placebo for one month, and the group that had placebo in the first treatment phase will take melatonin for one month. A last polysomnography will be recorded after the second treatment phase.

The other medications (antiepileptic drugs) taken by the patients before the trial will not be modified.

ELIGIBILITY:
Inclusion Criteria:

* Lennox-Gastaut syndrome (based on ILAE classification, 1989)
* light mental retardation (QI 50-69)
* french mother tongue
* having someone helping the patient (parent and/or referent educator)
* informed consent have been given by the patient / guardian
* absence of concomitant evolutive affection or associated sleep pathologies
* collaboration of the patient, ability to complete all aspects of the trial.

Exclusion Criteria:

* epileptic syndrome other than Lennox-Gastaut, other neurologic and/or psychiatric disease
* moderate to severe mental retardation (QI < 50)
* psychiatric disease that could interfere with the diagnostic procedure
* specific sleep disorder (anamnestic and diagnosed on the polygraphic record), for example: sleep apnea syndrome, narcolepsy, restless legs syndrome, periodic legs movements, etc...

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
diminution of at least 50% of the nocturnal interictal discharges and tonic seizures with the melatonin treatment | assessed after 1 month and 2.5 months
  The patients will have three polysomnographic recording: at the baseline, one month after initiating the treatment (melatonin or placebo) and one month after the cross-over phase. The number of tonic seizure and if interictal discharges will be assessed.
  The primary outcome measure is a diminution of > 50% of the seizures/interictal discharges with the melatonin treatment.

SECONDARY OUTCOMES:
augmentation of at least 15% of the amount of deep slow sleep with the melatonin treatment | assessed after 1 month and 2.5 months.
  The structure of sleep will be measured with the polysomnography (at baseline, after 1 month and after 2.5 months.
  The outcome measure is an augmentation of at least 15% of the deep slow sleep.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni B. Foletti, MD, MER, Principal Investigator — Institution de Lavigny
Locations (1):
- Institution de Lavigny, Lavigny, Canton of Vaud, Switzerland